CLINICAL TRIAL: NCT03409757
Title: Velphoro and Impact on the Oral Cavity and Gut Microbiome
Acronym: MicrobiomEisen
Status: Terminated | Type: Observational
Why Stopped: Insufficient Patient Recruitment
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-058
Record Dates: First submitted 2017-12-05; First posted 2018-01-24 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Hyperphosphatemia
Keywords: microbiome
MeSH Terms: conditions — Hyperphosphatemia | interventions — sucroferric oxyhydroxide; Transdermal Patch; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gingival biofilm, saliva and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hemodialysis patients with hyperphosphatemia: * dental investigation and two sample collections of saliva, gingival biofilm (plaque) and stool
  * Velphoro® medication
  Interventions: Drug: Velphoro; Other: saliva collection; Other: Supragingival biofilm collection; Other: stool collection; Other: blood collection
- control group: - dental investigation and two sample collections of saliva, gingival biofilm (plaque) and stool
  Interventions: Other: saliva collection; Other: Supragingival biofilm collection; Other: stool collection

INTERVENTIONS:
Drug: Velphoro — 4 weeks
  Other Names: Sucroferric oxyhydroxide
  Groups: hemodialysis patients with hyperphosphatemia
Other: saliva collection — 2 samples
Other: Supragingival biofilm collection — 2 samples
  Other Names: plaque
Other: stool collection — 2 samples
Other: blood collection — 2 samples
  Groups: hemodialysis patients with hyperphosphatemia

SUMMARY:
This pilot study will be carried out to determine if the regular intake of iron-based Velphoro® by hyperphosphatemia patients influences the microbiome in the oral cavity and/or the gut.

DETAILED DESCRIPTION:
The aim of this study is to investigate potential changes in the microbiome of the oral cavity and/or gut in patients with hyperphosphatemia following Velphoro® intake for one month. The principal intention of this study is to assess consequences of Velphoro® medication beyond phosphate control. Adherence to the drug might be compromised by e.g. staining of teeth and biofilm after chewing the product more than recommended. Most likely this is a cosmetic problem only and easy to solve by optimizing oral hygiene. The increased level of iron may have an effect on the gut microbiome which could lead to mild diarrhoea. However, the present study will assess, whether the microbiome both oral and gut changes significantly due to some iron bio-availability, although this is expected to be low with sucroferric oxyhydroxide.

The ultimate goal is to improve patient adherence to the drug and to resolve potential safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from hyperphosphatemia
* Current treatment with a stable dose of a non-iron containing phosphate binder,
* No or only parenteral iron application
* Age of ≥ 18 years
* Written informed consent prior to study participation
* The subject is willing and able to follow the procedures outlined in the protocol

Control group:

* Normal renal function
* No hyperphosphatemia
* Age- and sex-matched and oral disease status-matched (dental caries and periodontal disease) in comparison to the hyperphosphatemia group
* Written informed consent prior to study participation
* The subject is willing and able to follow the procedures outlined in the protocol

Exclusion Criteria:

* Age less than 18 years
* Currently on oral iron application
* Antibiotic treatment within the last two months
* Severe medical events within the last three months
* Planned surgery for the duration of the sampling
* Acute/chronic gastrointestinal infections
* Smokers
* Oral candidiasis
* Oral cancer
* Pregnant and lactating females
* Haemochromatosis history
* Committed to an institution by legal or regulatory order
* Participation in a parallel interventional clinical trial
* Receipt of an investigational drug within 30 days prior to inclusion into this study
* The subject is mentally or legally incapacitated

Only for the patient group:

* Never got any phosphate binder
* Allergy to Velphoro®
* Celiac disease or any other chronic inflammatory bowel disease
* Previous major surgery in the gastrointestinal tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hemodialysis patients suffering from hyperphosphatemia and healthy volunteers from the clinical routine in the Department of Operative Dentistry, Periodontology and Preventive Dentistry at the university hospital RWTH Aachen
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
change in relative abundances of iron depending bacterial species within the microbiome from before Velphoro medication to afterwards | 4 weeks

SECONDARY OUTCOMES:
Change of distribution of bacterial species within the microbiome from baseline to after Velphoro medication | 4 weeks
  via diversity measure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of RWTH Aachen, Department of Medicine II, Aachen, Germany